CLINICAL TRIAL: NCT06341790
Title: Effect of Consumption of Millets Based Diet on, Clinical Characteristics, Metabolic Profile, and Gut Microbiome in Patients With Non-alcoholic Fatty Liver Disease
Brief Title: Effect of Consumption of Millet Diet in Patients With NAFLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NAFLD-02
Record Dates: First submitted 2024-03-04; First posted 2024-04-02 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-03

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A-Normal diet (No Intervention): patients are advised normal diet for NAFLD
- Group b-Millet Diet (Experimental): Patients are given millets based diet (jowar)
  Interventions: Other: jowar based products

INTERVENTIONS:
Other: jowar based products — jowar based products like jowar flakes, jowar aata, jowar vermicelli is given to the intervention group
  Arms: Group b-Millet Diet

SUMMARY:
With NAFLD fast rising its ranks in becoming a major non communicable disease in India and across the globe, this study aims at primary prevention of the condition. NAFLD is a spectrum of diseases characterised by the deposition of fat within hepatocytes and is a precursor of liver inflammation. Global estimates peg the prevalence to be around 30 to 40%, but there are not many studies which have documented the prevalence in India. With the epidemiological transition, the cases of NAFLD are also on a rise as metabolic syndrome is an important risk factor.

It is apparent that the westernized way of our lifestyle especially the junk food culture comprising of super portions of loads of calories, sugars and salts is the main driver of this nutritional pandemic. The traditional diets in India were rich in fruits and vegetables, low in simple carbohydrates and high in fibre. Cereals are the main source of calories in any diet, forming the base of the food pyramid. Managing our cereals from being refined to the more complex ones being rich in fibre, protein and good quality fat could be a major player in the whole game of dietary modifications not just therapeutically but also prophylactically. Hence our therapeutic focus should be in increasing the consumption of cereals that are not only high in fibre, low in carbohydrates but also that have the potential to modulate the intestinal bacterial ecology to a more favourable type thus helping in intensifying the effects of overall dietary modifications.

Gut microbiota is currently explored for its role in NAFLD and there are gaps in knowledge which preclude having therapeutic strategies through its modulation. Millets, which were once considered to be poor man's diet are now becoming a part of the plate more frequently, especially for its unique nutritive content, with increased fiber, low carbohydrates, high protein and good quality fats. The processing methods may alter glycemic responses. Thus, the present study is proposed to look into the effect of millet based diets in reduction of hepatic steatosis and the resultant alterations in the gut microbiota .

DETAILED DESCRIPTION:
a) Aim and Objective - Primary Objectives

• To study the effect of millets based diet on hepatic steatosis in patients with NAFLD

Secondary Objective:

* To study the effect of millets based diet on metabolic features like blood sugar levels, HbA1C, Insulin resistance, Lipid profile, and liver transaminases in patients with NAFLD.
* To study the effect of millets based diet on body composition in patients with NAFLD
* To study the effect of millets based diet on the profile of gut microbiota in patients with NAFLD (b) Methodology:

  * Study population: Out patients of departments of Hepatology and Clinical Nutrition, Institute of Liver and Biliary Sciences, New Delhi.
  * Study design: Randomized Controlled Trial - an open label study
  * Study Protocol: Newly diagnosed patients with non-alcoholic fatty liver (NAFL) attending the outpatient departments of Hepatology and Clinical Nutrition would be screened for eligibility for randomization into the study as per the inclusion and exclusion criteria. Thereafter the eligible patients would be randomized into the two groups - the control group (standard diet group) and the intervention group (Millets based diet group). All the patients would undergo a detailed clinical evaluation. Information would be collected regarding the onset and duration of symptoms, etiology, and severity of disease, other baseline clinical features, routine biochemical and hematological investigations, nutritional assessment. All the patients would be followed up at regular intervals in the OPD. Repeat assessment of all the parameters would be done at the end of intervention period of three months also.
  * Study Duration: 2 yrs
  * Follow up period: 3 months
  * Inclusion Criteria:
  * Recently diagnosed consenting adults with NAFL (steatotosis) of any grade with or without features of metabolic syndrome, diagnosed on the basis of ultrasound and /or liver transient eleastography (controlled attenuation parameter; CAP >250).
  * Age 18-60 years
  * Exclusion Criteria:
  * Pregnant & lactating women
  * Age <18 and >60 years
  * Individuals who had been hospitalised with complications of Diabetes mellitus, Chronic Kidney disease, Hypertension in the previous 6 months
  * Those with intake of antibiotics within last month
  * Seriously ill and bed ridden patients
  * Patients with viral hepatitis
  * Patients with significant alcohol consumption (regular consumption of > 10g per day for females and > 20g/d in males),
  * Patients having chronic inflammatory bowel disease or any chronic and autoimmune diseases will be excluded
  * Patients with NAFLD with associated hypertriglyceridemia that requires administration of statins.
  * Sample size with justification:
  * As there is no literature available on the direct effect of Millets based diet on NAFLD, hence the present study would be a proof of concept study. The total sample size planned is 60 patients with NAFLD i.e. 30 patients each in the control and intervention group.
  * Intervention: Nutritional Intervention with Millets including Ragi Flakes; Pearl Millet Flakes; Multi Millet Roti; Foxtail Millet Rice.
  * Intervention Groups:Control Group A (Standard Diet Group): This group would receive standard nutritional counselling with customized diet providing 20-25 Kcal/Kg and 1.0 gm protein/kg ideal body wt/day. 15-20% of the total calories as proteins, 50-60% of carbohydrates (Main Source: Wheat, Rice, Oats) and 25-30% of fats. Diet would be planned keeping in mind the individual food habits and choices. This group would not receive any nutritional supplement other than the prescribed diet.
  * Intervention Group B (Millets Diet Group): This group would receive standard nutritional counselling, customized diet providing 20-25 Kcal/Kg and 1.0 gm protein/kg ideal body wt/day. 15-20% of the total calories as proteins, 50-60% of carbohydrates (Main Source: Pearl millet flakes/Foxtail millet rice/multi millet roti) and 20-25% of fats. Diet would be planned keeping in mind the individual food habits and choices. This group would not receive any nutritional supplement other than the prescribed diet.
  * Physical activity recommendations: Brisk walking on a treadmill (at a speed 5-6 Kmph for 45 minutes) OR 5000 steps per day by pedometer counting
  * Duration of Intervention: Diets would be given for a period of three months.
  * Stopping rule for intervention:
  * Temporary Stopping Rules during the Study

    1. Non-compliance
    2. Allergic response to millets intervention
    3. Voluntary withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* - Recently diagnosed consenting adults with NAFL (steatotosis) of any grade with or without features of metabolic syndrome, diagnosed on the basis of ultrasound and /or liver transient eleastography (controlled attenuation parameter; CAP >250).
* Age 18-60 years

Exclusion Criteria:

* - Pregnant & lactating women
* Age <18 and >60 years
* Individuals who had been hospitalised with complications of Diabetes mellitus, Chronic Kidney disease, Hypertension in the previous 6 months
* Those with intake of antibiotics within last month
* Seriously ill and bed ridden patients
* Patients with viral hepatitis
* Patients with significant alcohol consumption (regular consumption of > 10g per day for females and > 20g/d in males),
* Patients having chronic inflammatory bowel disease or any chronic and autoimmune diseases will be excluded
* Patients with NAFLD with associated hypertriglyceridemia that requires administration of statins.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2026-07-05 (Estimated); Study Completion 2026-07-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of hepatic steatosis in NAFLD patients | 3months
  Change in hepatic steatosis as assessed by fibroscan, ultrasound (change in the CAP, LSM)

SECONDARY OUTCOMES:
Assessment of blood sugar | 3months
  Change in blood sugar as assessed by blood fasting glucose, serum insulin & HbA1c
Assessment of lipid function | 3 months
  Change in lipid parameters as assessed by blood lipid profile test
Assessment of liver transaminases | 3 months
  Change in liver enzymes as assessed by liver function tests
Assessment of body composition | 3 months
  Change in Nutritional status will be assessed using bioelectrical impedence analysis
Assessment of Gut Microbiota | 3months
  Change in gut microbiota will be assessed using 16S dNA extraction

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jaya Joy Benajmin, Phd, Principal Investigator — Associate Professor, Clinical Nutrition at the Institute of Liver and Biliary Sciences (ILBS)
Locations (1):
- ILBS, New Delhi, India

IPD SHARING:
Plan to Share IPD: No